CLINICAL TRIAL: NCT01559389
Title: Incontinence & Intimate Partners: Assessing the Contribution of Treatment
Acronym: IIMPACT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Loyola University (Other)
Collaborators: Astellas Pharma US, Inc. (Industry)
Responsible Party: Principal Investigator, Elizabeth Mueller, Associate Professor, Loyola University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 203952
Record Dates: First submitted 2012-03-15; First posted 2012-03-21 (Estimated); Results first posted 2019-12-02 (Actual); Last update posted 2019-12-02 (Actual); Status verified 2019-11

CONDITIONS: Urge Urinary Incontinence
Keywords: Urge Urinary Incontinence; Vesicare; Urinary Incontinence; Sexual function; solifenacin
MeSH Terms: conditions — Urinary Incontinence, Urge; Urinary Incontinence | interventions — Solifenacin Succinate

STUDY DESIGN:
Intervention Model Description: Women presenting with UUI symptoms will receive up to 16 weeks of solifenacin.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Female Partners (Experimental): This arm comprises female partners who receive up to 16 weeks of solifenacin treatment for their UUI symptoms
  Interventions: Drug: Solifenacin
- Male Partners (No Intervention): This arm comprises healthy male partners

INTERVENTIONS:
Drug: Solifenacin — Women presenting with UUI symptoms receive 5 to 10 milligrams (mg) of daily solifenacin for up to 16 weeks
  Other Names: Vesicare
  Arms: Female Partners

SUMMARY:
Urge urinary incontinence (UUI) is a socially debilitating disease due to its inherently unpredictable nature and sometimes large volumes of urine loss. Women with UUI may experience anxiety over public episodes of incontinence and concerns about odor and, as a result, isolate themselves socially. This isolation affects both partners in the relationship and may be a source of discord. The impact of UUI also moves into personal relationships where fears or actual episodes of incontinence during physical intimacy, including but limited to intercourse, may result in limited interactions and changes in the relationship satisfaction for both partners. Few studies have examined the role of urinary incontinence, particularly UUI, in the dynamics of an intimate partner relationship and none have evaluated the impact of successful UUI treatment.

The long-term goal of our research is to understand the social and emotional impact of pelvic floor disorders, particularly UUI, on the well-being of an intimate relationship. Ultimately, we aim to evaluate the role that successful treatment plays in the alleviation of discord in intimate partner relationships that are affected by UUI and other pelvic floor disorders.

Our objective for this proposal is to characterize, using validated, quantifiable methods the quality of the relationship in couples affected by UUI and to identify the role that treatment plays in improving this relationship. Our central hypothesis is that UUI has a negative impact upon the emotional and physical well-being of a relationship and that effective treatment will result in improvement in areas of the relationship that have been detrimentally affected by UUI. Our rationale for this study is that an understanding of UUI in the context of a couple, particularly from the perspective of the male partner, will improve our ability to holistically treat UUI, thus improving patient outcomes and satisfaction.

DETAILED DESCRIPTION:
Chronic illness places emotional, physical, and financial burdens upon both the patient and her partner and can be a significant source of stress in a relationship. The symptoms of UUI inherently pose greater social challenges than those faced by women other forms of pelvic floor disorders. For example, women with UUI may avoid social situations due to fear of having an accident or may be reluctant to participate in activities during which it may be difficult to find a bathroom. The resulting social isolation impacts both members of the dyad and may serve as a source of relationship discord. Changes in sexual function and perceived intimacy, including non-intercourse intimacy, as well as communication may be new sources of stress in a previously healthy relationship or may serve to amplify pre-existing relationship problems.

Sexual function is another area in which UUI may cause a negative impact. Studies of coital incontinence among incontinent clinic populations report prevalence ranging from 10%-56% with a median of 22%. The prevalence of coital incontinence may be related to the type of incontinence as well as the severity of symptoms. Stress incontinence has been associated with leakage of urine during intercourse, while detrusor instability and urge incontinence have been correlated with leakage during orgasm. A cross-sectional study of women with UUI and urinary incontinence found that among women reporting low sexual desire, stress incontinence was common (47%), while 46% of women reporting orgasmic phase dysfunction reported symptoms of urge incontinence. Qualitative data corroborates the negative impact of UUI on dyadic and sexual relations.

Another mechanism by which UUI may affect satisfaction with dyadic relations is through depressive symptomatology. Urinary incontinence is associated with a decrease in overall health-related quality of life and is positively correlated with depression, anxiety, and stress. Studies of other chronic illnesses demonstrate a correlation between the patient's level of depression and that of their spouse; level of depression shows an inverse relationship with degree of satisfaction with the relationship.

One of the two studies in the published literature that use quantitative methods to evaluate the impact of urodynamic stress incontinence and detrusor overactivity on the marital relationship concluded that both sexual function and marital relationships are negatively affected by incontinence. This study, like others, is based upon the perspective of the female partner. A recent study of Swedish women with urinary incontinence and urgency is the only study which includes the perspective of the male partner to examine the impact of UUI on the relationship. It concludes that, "Female urinary incontinence, urgency and frequency significantly impair the quality of life in both younger and older women, and also have negative effects on the partner relationship and the partner's life".

The perspective of intimate partners of women with UUI and other forms of PFD is largely missing from the literature. Any analysis of the role of UUI in intimate partner relationships is incomplete without this perspective.

ELIGIBILITY:
Healthy male partners may volunteer to participate in this study along with their affected female partners. There are no inclusion or exclusion criteria for male partners.

For affected female participants, the following inclusion criteria apply:

* Age ≥ 18 years
* In a relationship with a male partner for at least 3 months
* Not pregnant or planning to become pregnant
* Have a diagnosis of UUI or Mixed Urinary Incontinence (MUI) that is urge predominant based on a 3 day voiding diary
* Are interested in medical management of their symptoms
* Are candidates for solifenacin
* Are able to provide informed consent
* Are able to complete written questionnaires.

For affected female partners, the following exclusion criteria apply:

* Post Voided Residual (PVR) > 200 ml at the initial visit
* History of a significant outflow obstruction
* History of persistent/recurrent Urinary Tract Infection (UTI)
* History of bladder stones
* History of a diagnosis of chronic interstitial cystitis
* History of pelvic irradiation
* Current pelvic malignancy
* Narrow angle glaucoma
* Urinary or gastric retention
* Current use of a tricyclic antidepressant
* A neurologic diagnosis that could affect bladder function
* History of chronic pelvic pain
* Active psychotic disorder
* Male partner does not speak English
* Declines permission for the study team to recruit their male partner for the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 138 (Actual)
Dates: Start 2012-03-09 (Actual); Primary Completion 2017-06-29 (Actual); Study Completion 2017-06-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Meuller, MD, Principal Investigator — Loyola University
Locations (1):
- Loyola University Medical Center, Maywood, Illinois, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan to share individual participant data

REFERENCES:
- [Background] Shaw C. A systematic review of the literature on the prevalence of sexual impairment in women with urinary incontinence and the prevalence of urinary leakage during sexual activity. Eur Urol. 2002 Nov;42(5):432-40. doi: 10.1016/s0302-2838(02)00401-3. PMID 12429150
- [Background] Hilton P. Urinary incontinence during sexual intercourse: a common, but rarely volunteered, symptom. Br J Obstet Gynaecol. 1988 Apr;95(4):377-81. doi: 10.1111/j.1471-0528.1988.tb06609.x. PMID 3382610
- [Background] Salonia A, Zanni G, Nappi RE, Briganti A, Deho F, Fabbri F, Colombo R, Guazzoni G, Di Girolamo V, Rigatti P, Montorsi F. Sexual dysfunction is common in women with lower urinary tract symptoms and urinary incontinence: results of a cross-sectional study. Eur Urol. 2004 May;45(5):642-8; discussion 648. doi: 10.1016/j.eururo.2003.11.023. PMID 15082208
- [Background] Coyne KS, Matza LS, Brewster-Jordan J. "We have to stop again?!": The impact of overactive bladder on family members. Neurourol Urodyn. 2009;28(8):969-75. doi: 10.1002/nau.20705. PMID 19301410
- [Background] Bovbjerg VE, Trowbridge ER, Barber MD, Martirosian TE, Steers WD, Hullfish KL. Patient-centered treatment goals for pelvic floor disorders: association with quality-of-life and patient satisfaction. Am J Obstet Gynecol. 2009 May;200(5):568.e1-6. doi: 10.1016/j.ajog.2008.11.020. Epub 2009 Feb 23. PMID 19236871
- [Background] Coyne KS, Wein AJ, Tubaro A, Sexton CC, Thompson CL, Kopp ZS, Aiyer LP. The burden of lower urinary tract symptoms: evaluating the effect of LUTS on health-related quality of life, anxiety and depression: EpiLUTS. BJU Int. 2009 Apr;103 Suppl 3:4-11. doi: 10.1111/j.1464-410X.2009.08371.x. PMID 19302497
- [Background] Litman HJ, Steers WD, Wei JT, Kupelian V, Link CL, McKinlay JB; Boston Area Community Health Survey Investigators. Relationship of lifestyle and clinical factors to lower urinary tract symptoms: results from Boston Area Community Health survey. Urology. 2007 Nov;70(5):916-21. doi: 10.1016/j.urology.2007.06.1117. Epub 2007 Oct 24. PMID 17919693
- [Background] Daneker B, Kimmel PL, Ranich T, Peterson RA. Depression and marital dissatisfaction in patients with end-stage renal disease and in their spouses. Am J Kidney Dis. 2001 Oct;38(4):839-46. doi: 10.1053/ajkd.2001.27704. PMID 11576888
- [Background] Yip SK, Chan A, Pang S, Leung P, Tang C, Shek D, Chung T. The impact of urodynamic stress incontinence and detrusor overactivity on marital relationship and sexual function. Am J Obstet Gynecol. 2003 May;188(5):1244-8. doi: 10.1067/mob.2003.273. PMID 12748492
- [Background] Nilsson M, Lalos A, Lalos O. The impact of female urinary incontinence and urgency on quality of life and partner relationship. Neurourol Urodyn. 2009;28(8):976-81. doi: 10.1002/nau.20709. PMID 19229955
- [Background] Barber MD, Walters MD, Bump RC. Short forms of two condition-specific quality-of-life questionnaires for women with pelvic floor disorders (PFDI-20 and PFIQ-7). Am J Obstet Gynecol. 2005 Jul;193(1):103-13. doi: 10.1016/j.ajog.2004.12.025. PMID 16021067
- [Background] Herzog AR, Diokno AC, Brown MB, Normolle DP, Brock BM. Two-year incidence, remission, and change patterns of urinary incontinence in noninstitutionalized older adults. J Gerontol. 1990 Mar;45(2):M67-74. doi: 10.1093/geronj/45.2.m67. PMID 2313045
- [Background] Rogers RG, Coates KW, Kammerer-Doak D, Khalsa S, Qualls C. A short form of the Pelvic Organ Prolapse/Urinary Incontinence Sexual Questionnaire (PISQ-12). Int Urogynecol J Pelvic Floor Dysfunct. 2003 Aug;14(3):164-8; discussion 168. doi: 10.1007/s00192-003-1063-2. Epub 2003 Jul 25. PMID 12955337
- [Background] Rust J, Golombok S. The Golombok-Rust Inventory of Sexual Satisfaction (GRISS). Br J Clin Psychol. 1985 Feb;24 ( Pt 1):63-4. doi: 10.1111/j.2044-8260.1985.tb01314.x. PMID 3971070
- [Background] Spanier GB. The measurement of marital quality. J Sex Marital Ther. 1979 Fall;5(3):288-300. doi: 10.1080/00926237908403734. PMID 513146
- [Background] Johnson SM, Greenberg LS. Differential effects of experiential and problem-solving interventions in resolving marital conflict. J Consult Clin Psychol. 1985 Apr;53(2):175-84. doi: 10.1037//0022-006x.53.2.175. No abstract available. PMID 3998245
- [Background] Jacobson NS. A component analysis of behavioral marital therapy: the relative effectiveness of behavior exchange and communication/problem-solving training. J Consult Clin Psychol. 1984 Apr;52(2):295-305. doi: 10.1037//0022-006x.52.2.295. No abstract available. PMID 6715653
- [Background] Jacobson NS, Follette WC, McDonald DW. Reactivity to positive and negative behavior in distressed and nondistressed married couples. J Consult Clin Psychol. 1982 Oct;50(5):706-14. doi: 10.1037//0022-006x.50.5.706. No abstract available. PMID 7142544
- [Background] Nathan EP, Joanning HH. Enhancing marital sexuality: an evaluation of a program for the sexual enrichment of normal couples. J Sex Marital Ther. 1985 Fall;11(3):157-64. doi: 10.1080/00926238508405441. PMID 4068043

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited from March 2012 through July 2016 (52 months) from the Division of Female Pelvic Medicine & Reconstructive Surgery at Loyola University Medical Center.
Groups:
- Females With UUI: This arm comprises female partners who receive up to 16 weeks of solifenacin treatment for their UUI symptoms
- Male Partners: This arm comprises the healthy male partners of the female participants
Period: Overall Study
Arm/Group | Females With UUI | Male Partners
Started | 69 | 69
Completed | 49 | 49
Not Completed | 20 | 20
Not completed — Withdrawal by Subject | 20 | 20

BASELINE CHARACTERISTICS:
Population: The baseline analysis population comprises the 49 of 69 couples who enrolled and completed the GRISS questionnaire at both timepoints.
Groups:
- Females With UUI: This arm comprises females who receive up to 16 weeks of solifenacin treatment for their UUI symptoms
- Total: Total of all reporting groups
Arm/Group | Females With UUI | Male Partners | Total
Number analyzed (Participants) | 49 | 49 | 98
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 49 | 49 | 98
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 49 | 0 | 49
  Male | 0 | 49 | 49
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 37 | 36 | 73
  Black | 8 | 8 | 16
  Asian | 0 | 1 | 1
  Hispanic | 4 | 3 | 7
  Other | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 49 | 49 | 98
Marital Status [Count of Participants; unit: Participants]
  Married | 42 | 42 | 84
  Divorced | 3 | 1 | 4
  Single | 4 | 6 | 10
Education [Count of Participants; unit: Participants] — Population: Information on education is only collected for female participants
  Participants
    number analyzed (Participants) | 49 | 0 | 49
    High school or less | 19 | 0 | 19
    At least some college | 29 | 0 | 29
    Not reported | 1 | 0 | 1
Years with Partner [Count of Participants; unit: Participants]
  Fewer than 30 years | 24 | 23 | 47
  30 or more years | 25 | 26 | 51
Body Mass Index [Count of Participants; unit: Participants] — Population: Information on body mass index is only collected for female participants
  Participants
    number analyzed (Participants) | 49 | 0 | 49
    Less than 30 kg/m^2 | 19 |  | 19
    30 kg/m^2 or more | 30 |  | 30
Menstrual Cycle [Count of Participants; unit: Participants] — Population: Information on menopause is only collected for female participants
  Participants
    number analyzed (Participants) | 49 | 0 | 49
    Pre-menopausal | 9 | 0 | 9
    Post-menopausal | 38 | 0 | 38
    Not certain | 2 | 0 | 2
Vaginal Parity [Count of Participants; unit: Participants] — Population: Information on parity is only collected for female participants
  Participants
    number analyzed (Participants) | 49 | 0 | 49
    0-1 births | 8 | 0 | 8
    2 births | 20 | 0 | 20
    3 births | 10 | 0 | 10
    4-6 births | 11 | 0 | 11
Prior Surgery [Count of Participants; unit: Participants] — Population: Information on prior surgery is only collected for female participants
  Participants
    number analyzed (Participants) | 49 | 0 | 49
    Yes | 27 |  | 27
    No | 22 |  | 22
Prior Treatments for Overactive Bladder Syndrome [Count of Participants; unit: Participants] — Population: Information on prior treatments for Overactive Bladder Syndrome is only collected for female participants
  Participants
    number analyzed (Participants) | 49 | 0 | 49
    Yes | 19 |  | 19
    No | 30 |  | 30
Prior Treatment for Pelvic Floor Disorders [Count of Participants; unit: Participants] — Population: Measure Analysis Population Description: Information on prior treatments for pelvic floor disorders is only collected for female participants
  Participants
    number analyzed (Participants) | 49 | 0 | 49
    Yes | 20 |  | 20
    No | 29 |  | 29
General Health [Count of Participants; unit: Participants]
  Excellent | 4 | 8 | 12
  Very Good | 10 | 16 | 26
  Good | 25 | 16 | 41
  Fair | 8 | 8 | 16
  Poor | 2 | 1 | 3
Medical History [Count of Participants; unit: Participants] — Population: Information on hypertension, erectile dysfunction, arthritis, diabetes, cancer, heart disease, and depression is only collected for male participants
  Participants
    Hypertension: number analyzed (Participants) | 0 | 49 | 49
    Hypertension | 0 | 16 | 16
    Erectile dysfunction: number analyzed (Participants) | 0 | 49 | 49
    Erectile dysfunction | 0 | 13 | 13
    Arthritis: number analyzed (Participants) | 0 | 49 | 49
    Arthritis | 0 | 13 | 13
    Diabetes: number analyzed (Participants) | 0 | 49 | 49
    Diabetes | 0 | 9 | 9
    Cancer: number analyzed (Participants) | 0 | 49 | 49
    Cancer | 0 | 9 | 9
    Heart disease: number analyzed (Participants) | 0 | 49 | 49
    Heart disease | 0 | 6 | 6
    Depression: number analyzed (Participants) | 0 | 49 | 49
    Depression | 0 | 6 | 6
Currently Sexually Active [Count of Participants; unit: Participants] — Population: Information on current sexual activity is only collected for male participants
  Participants
    number analyzed (Participants) | 0 | 49 | 49
    Yes |  | 36 | 36
    No |  | 13 | 13

OUTCOME MEASURES:

1. Primary Outcome: Baseline Sexual Satisfaction Between Matched Female and Male Partners
Description: Prior to beginning treatment with solifenacin, females presenting with UUI complete the Golombok Rust Inventory of Sexual Satisfaction (GRISS). Their male partners also complete the GRISS at the baseline visit. The GRISS is a 28-item self-administered questionnaire that assess the quality of the sexual relationship of a heterosexual couple. Scores range from 0 to 10 with higher scores indicating greater sexual dysfunction.
Time Frame: 0 Weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Females With UUI | Male Partners
Number analyzed (Participants) | 49 | 49
score on a scale | 4.2 (2.3) | 4.8 (2.4)
Statistical Analysis 1: Comparison: Females With UUI vs Male Partners; The null hypothesis is that there is no difference in the overall GRISS score between females with UUI and their male partners; Test type: Superiority; p = .16, t-test, 2 sided — P-values less than 0.05 were considered statistically significant; The method was a paired t-test; Mean Difference (Final Values) = -0.51, 95% CI 2-sided [-1.23 to 0.21], Standard Deviation 2.50

2. Secondary Outcome: Change in Overall Sexual Satisfaction Among Females
Description: Females presenting with UUI complete the Golombok Rust Inventory of Sexual Satisfaction (GRISS) at baseline (0 weeks) and after 12-16 weeks of treatment with solifenacin. For this outcome, the baseline score is subtracted from the follow-up score and this change score is compared between those who respond and do not respond to treatment with solifenacin. The GRISS is a 28-item self-administered questionnaire that assess the quality of the sexual relationship of a heterosexual couple. Scores range from 0 to 10 with higher scores indicating greater sexual dysfunction.
Time Frame: Baseline and 12-16 weeks
Population: The analysis population comprises 49 female participants who received up to 16 weeks of solifenacin for the treatment of UUI symptoms
Measure: Median (Inter-Quartile Range); unit: score on a scale
Groups:
- Responder: This arm comprises female participants who respond to solifenacin treatment for their UUI symptoms. Response to treatment comprises those who rate their Global Impression of Improvement (GII) as "a little better", "much better", or "very much better"
- Non-Responder: This arm comprises female participants who do not respond to solifenacin treatment for their UUI symptoms. Non-response to treatment is defined as those who rate their Global Impression of Improvement (GII) as "no change", "a little worse", "much worse", and "very much worse".
Arm/Group | Responder | Non-Responder
Number analyzed (Participants) | 14 | 35
score on a scale | -0.5 [-1 to 0] | 0 [0 to 1]
Statistical Analysis 1: Comparison: Responder vs Non-Responder; The null hypothesis is that there is no difference in the overall GRISS change score between those who respond and do not respond to treatment with solifenacin; Test type: Superiority; p = .003, Wilcoxon (Mann-Whitney); Exact test; z-score = 2.97 — The z-score is a standardized Wilcoxon statistic. In this study, z-scores with an absolute value exceeding 1.96 indicate a significant difference in the GRISS change score between responders and non-responders of solifenacin treatment

3. Secondary Outcome: Change in Overall Sexual Satisfaction Among Healthy Male Partners
Description: Healthy male partners of female participants complete the Golombok Rust Inventory of Sexual Satisfaction (GRISS) survey. For this outcome, their baseline score is subtracted from their follow-up score which is collected after their female partner completes approximately 12-16 weeks of solifenacin treatment for UUI symptoms. This change score is compared between male partners of female participants who respond to solifenacin versus male partners of female participants who do not respond to solifenacin. The GRISS is a 28-item self-administered questionnaire that assess the quality of the sexual relationship of a heterosexual couple. Scores range from 0 to 10 with higher scores indicating greater sexual dysfunction.
Time Frame: Baseline and 12-16 weeks
Population: The analysis population comprises the 49 male partners of the female participants who received up to 16 weeks of solifenacin for the treatment of UUI symptoms
Measure: Median (Inter-Quartile Range); unit: score on a scale
Groups:
- Male Partners of Female Responders: This arm comprises the male partners of female participants who respond to solifenacin treatment for their UUI symptoms
- Male Partners of Female Non-Responders: This arm comprises the male partners of female participants who do not respond to solifenacin treatment for their UUI symptoms
Arm/Group | Male Partners of Female Responders | Male Partners of Female Non-Responders
Number analyzed (Participants) | 14 | 35
score on a scale | 0 [0 to 0] | 0 [-1 to 0]
Statistical Analysis 1: Comparison: Male Partners of Female Responders vs Male Partners of Female Non-Responders; The null hypothesis is that there is no difference in the overall GRISS change score between male partners of female participants who respond to solifenacin and male partners of female participants who do not respond to solifenacin; Test type: Superiority; p = .37, Wilcoxon (Mann-Whitney); z-score = 0.89 — The z-score is a standardized Wilcoxon statistic. In this study, z-scores with an absolute value exceeding 1.96 indicate a significant difference in the GRISS change score between the two groups

ADVERSE EVENTS:
Time Frame: Adverse event data were collected for each female participant from March 2012 to June 2017 (i.e., 64 months)
Description: Male partners were not prescribed solifenacin and, consequently, were not at risk for adverse events. All-Cause Mortality, Serious, and Other (Not Including Serious) Adverse Events were not monitored/assessed for Male Partners.
Groups:
- Male Partners: This arm comprises the healthy male partners of the female participants. They were not prescribed solifenacin and, consequently, were not at risk for adverse events
Arm/Group | Females With UUI | Male Partners
All-Cause Mortality (participants affected / at risk) | 0/49 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/49 | 0/0
Other Adverse Events (participants affected / at risk) | 0/49 | 0/0

LIMITATIONS AND CAVEATS:
There are no limitations or caveats to report

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-06-01): https://cdn.clinicaltrials.gov/large-docs/89/NCT01559389/Prot_SAP_000.pdf